CLINICAL TRIAL: NCT02043821
Title: Maintenance Chemotherapy for Metastatic Colorectal Carcinoma
Brief Title: Maintenance Chemotherapy for Metastatic Colorectal Carcinoma and Biological Marker
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Dong Yan, Beijing Chao Yang Hospital, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20140116
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Other): Placebo 1250mg/m2 tablet by mouth every 12 hours for 14 days
  Interventions: Other: placebo
- Capecitabine (Experimental): Capecitabine 1250mg/m2 tablet by mouth every 12 hours for 14 days
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — 14days
  Arms: Capecitabine
Other: placebo — 14 days
  Arms: Placebo

SUMMARY:
Colorectal cancer patients with metastases (mCRC) at response under first-line chemotherapy are candidates for an convenient maintenance treatment.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common malignant tumors, with the morbidity of approximate 100 million cases per year. About 40% of patients present with metastatic (stage IV) colorectal cancer at the time of diagnosis, and about 25% of patients with local lesion will ultimately develop metastatic disease.Therefore, our study is designed to investigate that colorectal cancer patients with metastases (mCRC) at response under first-line chemotherapy are candidates for an convenient maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

- Age between 18 and 75 years Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1 histologically confirmed colorectal cancer with inoperable locally advanced or recurrent and/or metastatic disease Life expectancy of at least 3 months Intact organ function, including complete blood counts (CBC) showing normal values or any toxicity limited to grade 1 and blood chemistry (SMA) showing liver and renal functions < 1.5 upper normal limit (UNL).

Patients who achieved objective response or stable disease after 16-24 weeks first line chemotherapy Signed informed consent

Exclusion Criteria:

- Known hypersensitivity to capecitabine Concurrent any other cancer (except BCC or squamous cell carcinoma of skin). Inability to adhere to monthly visits to the oncology unit for evaluation. Presence of brain metastases. Previous radiotherapy to the only site of measurable disease. Evidence of severe or uncontrolled systemic disease No previous chemotherapy for metastatic disease Positive serum pregnancy test in women of childbearing potential unresolved bowel obstruction or malabsorption syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
DDC:Duration of Disease Control | 2 years
  progression-free survival of first-line chemotherapy with second-line chemotherapy

SECONDARY OUTCOMES:
OS:Overall Survival | 2 years
  measured from the initiation of chemotherapy to the date of the last follow-up or death
DCR:Disease Control Rate | 2 years
  This is defined as the occurrence of either a confirmed complete (CR),a partial response(PR)or stable disease(SD) as determined by the RECIST criteria from confirmed radiographic evaluations of target and non-target lesions.

OTHER OUTCOMES:
Safety | 2 years
  Adverse events and laboratory tests graded according to the NCI-CTC AE Version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Guangyu An, PhD, Study Director — Beijing Chao Yang Hospital